CLINICAL TRIAL: NCT02334163
Title: The Clinical Effects of Nitazoxanide in Hepatic Encephalopathy Patients: A Pilot Study
Brief Title: The Effects of Nitazoxanide in Hepatic Encephalopathy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Collaborators: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Asmaa Abdel Aziz ElRakaybi, Teaching assistant, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHCL400
Record Dates: First submitted 2015-01-06; First posted 2015-01-08 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Hepatic Encephalopathy
Keywords: Hepatic Encephalopathy; Nitazoxanide; Serum ammonia
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — nitazoxanide; Lactulose; Metronidazole; Rifaximin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nitazoxanide group (Experimental): 12 patients will receive the following for 7 days:
  * Oral lactulose
  * 500 mg nitazoxanide tablets twice daily
  Interventions: Drug: Nitazoxanide; Drug: Oral lactulose
- Metronidazole group (Active Comparator): 12 patients will receive the following for 7 days:
  * Oral lactulose
  * 250 mg metronidazole tablets every 8 hours
  Interventions: Drug: Oral lactulose; Drug: Metronidazole
- Rifaximine group (Active Comparator): 12 patients will receive the following for 7 days:
  * Oral lactulose
  * Two 200 mg rifaximine tablets every 8 hours
  Interventions: Drug: Oral lactulose; Drug: Rifaximine

INTERVENTIONS:
Drug: Nitazoxanide — 500 mg nitazoxanide tablets twice daily
  Arms: Nitazoxanide group
Drug: Oral lactulose — Oral lactulose (65%)
Drug: Metronidazole — 250 mg metronidazole tablets every 8 hours
  Arms: Metronidazole group
Drug: Rifaximine — Two 200 mg rifaximine tablets every 8 hours
  Arms: Rifaximine group

SUMMARY:
Evaluating the efficacy and safety of nitazoxanide in comparison to standard treatment in patients with grade II-III hepatic encephalopathy (HE). Also, Evaluating the effect of administering nitazoxanide on the improvement of patient's quality of life.

DETAILED DESCRIPTION:
Nitazoxanide (NTZ) is a thiazolide anti-infective with activity against anaerobic bacteria, protozoa and viruses. A pilot prospective study at the 2008 American Association for the Study of Liver Diseases meeting showing clinical improvement in HE among cirrhotic patients who received nitazoxanide and lactulose. Based on the excellent safety profile of NTZ, the present pilot study is conducted hopefully to prove the efficacy of nitazoxanide in treating patients experiencing HE grade II-III.

Study design:The study is Prospective, Randomized, Controlled, Open-Label, Pilot study.

Method: The study will include a total of 36 patients with grade II-III Hepatic Encephalopathy, and an informed consent will be obtained from every patient before being included.

All the patients will receive oral lactulose, plus either nitazoxanide, metronidazole or rifaximine.

A- All patients will be subjected to the following at baseline:

* Patient's full history
* Liver disease staging using Model for End stage Liver Disease (MELD) score
* Measurement of serum electrolytes (Na+, K+, Ca2+)

B- All patients will be subjected to the following at baseline and at the end of treatment:

* Measuring Blood ammonia level
* Measuring liver function tests (AST, Total bilirubin, international normalized ratio (INR), Serum albumin, prothrombin time (PT)), serum creatinine and complete blood count (CBC)
* Assessing severity of Hepatic Encephalopathy using Clinical Hepatic Encephalopathy Staging Scale (CHESS)

C- Monitoring tolerability up to 30 days after the last dose D- Assessment of quality of life using Chronic Liver Disease Questionnaire (CLDQ)

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients from 18 to 65 years.
* Patients with grade II-III Hepatic Encephalopathy.

Exclusion Criteria:

* Patients with active GIT bleeding.
* Patients with major psychiatric illness.
* Patients receiving benzodiazepines, narcotics, alcohol and marijuana.
* Patients with compromised renal or biliary functions.
* Patients known to have AIDS.
* Patients receiving medications highly bound to plasma proteins eg. Warfarin.
* Patients with known hypersensitivity to nitazoxanide.
* Pregnant or lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-02 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Evaluating the efficacy of nitazoxanide in improving mental status (calculating CHESS score) | 7 days
  evaluating the efficacy by measuring serum ammonia and calculating CHESS score at baseline and at end of treatment

SECONDARY OUTCOMES:
Evaluating the safety of nitazoxanide (estimation of treatment- related undesirable effects) | 37 days
  Evaluating the safety of nitazoxanide by estimation of treatment- related undesirable effects
Effect of nitazoxanide on patient's quality of life (CLDQ score) | 7 days
  Evaluating the effect on quality of life by calculating CLDQ score at baseline and at end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa A. Elrakaybi, Bachelor, Principal Investigator — Ain Shams University
Locations (1):
- Faculty of medicine, Ain Shams University, Cairo, Egypt